CLINICAL TRIAL: NCT05178212
Title: Characteristics and Outcomes of Patients With COVID-19-related Acute Respiratory Failure Treated With High-flow Nasal Oxygen and Awake-prone Position
Brief Title: Characteristics and Outcomes of Patients With COVID-19 Treated With HFNO and Prone Positioning
Acronym: AW-PP_Covid
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Collaborators: Hospital Aleman (Other); Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Mariano Esperatti, Mariano Esperatti, MD, PhD. Head of Section. Intensive Care Department. Hospital Privado de Comunidad. Mar del Plata. Argentina, Hospital Privado de Comunidad de Mar del Plata
Other Study IDs: AW-PP_Covid-19
Record Dates: First submitted 2021-12-23; First posted 2022-01-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2022-12

CONDITIONS: COVID-19; Respiratory Failure; Prone Position; Endotracheal Intubation; Mortality
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A subset of patients with COVID-19 develops acute respiratory failure and acute respiratory distress syndrome (ARDS) (1). The use of invasive mechanical ventilation for the treatment of these conditions is associated with high mortality rates (2,3). The use of high-flow nasal oxygen therapy (HFNO) and awake prone position (AW-PP) could to decrease the need for endotracheal intubation and other adverse clinical outcomes (4-6).

The aim of this study is to evaluate the clinical results of the simultaneous application of high-flow nasal oxygen therapy HFNO and awake-prone position in a cohort of patients with severe respiratory failure secondary to COVID-19 on relevant clinical outcomes, and to assess risk factors of treatment failure defined as requirement of invasive mechanical ventilation.

DETAILED DESCRIPTION:
Objective. To evaluate the clinical results of the simultaneous application of high-flow nasal oxygen therapy HFNO and awake-prone position in a cohort of patients with severe respiratory failure secondary to COVID-19 on relevant clinical outcomes, and to assess risk factors of treatment failure defined as requirement of invasive mechanical ventilation.

Design: Prospective multicenter cohort study conducted at 5 ICUs of 5 centers in Argentina. The Internal Review Board from the 5 centers approved the study including waived informed consent. The interventions carried out were part of the usual practice at each center and confidentiality of participants was guaranteed.

Population. Patients older than 18 years admitted to the ICU with a confirmed diagnosis of COVID-19 (real-time PCR) and receiving HFNO for at least 4 hours. Patients received HFNO when any of the following criteria were present: a) peripheral oxygen saturation (SpO2) < 92% with oxygen > 4 liters/minute; b) increased work of breathing with use of accessory respiratory muscles, and a respiratory rate > 30/min; c) partial pressure of oxygen /Fraction of inspired oxygen (PaO2/FiO2ratio) < 200 mmHg. Patients with respiratory failure secondary to a different etiology, decreased level of consciousness, presence of shock requiring vasopressors, immediate need for intubation, use of positive-pressure ventilation prior to HFNO, and with do-not intubate orders were excluded.

Procedures.Immediately after admission to the ICU, the inclusion criteria regarding oxygenation and/or work of breathing are checked. Then a high-flow nasal cannula sized according to the nares size is placed, and connected to a specific device for the provision of high-flow O2. The initial flow is 50-70 L/min, with the fraction of inspired oxygen (FiO2) necessary to obtain an SpO2 > 92%. No maximum FiO2 limits is established. Once therapy with HFNO is started, participants are encouraged and assisted by the health-care team to rotate from supine to prone position for as long as possible, taking breaks for personal hygiene and eating. No maximum time limits for prone position are established. Patients who tolerated HFNO for the next 4 hours are included in the study. These interventions are maintained during the study period until one of the following criteria was met: maintenance of SpO2 > 92% with FiO2 ≤ 40%, and flow ≤ 40 L/min for a period > 12 hours in the supine position; or endotracheal intubation. Analgesic drugs (opioids, paracetamol) or light sedation (dexmedetomidine) was allowed and indicated according to the criteria of the health-care team.

Variables and measurements. The following variables are collected: demographics (age, sex, body mass index [BMI]), comorbidities, severity scores upon ICU admission (APACHE II and SOFA), chronology of the disease (time from the onset of symptoms to hospital admission and ICU admission), vital signs, laboratory parameters, Respiratory rate Oxygenation index (ROX index) [7] , and chest computed tomography score (CT score) determined as the sum of lung involvement, ranging from 0 -no involvement- to 25 -maximum involvement [8].

Exposure: The main exposure of this study was awake prone positioning. The investigators will evaluate the number and proportion of patients who tolerate and cannot tolerate the prone position. For those who tolerate the prone position, the investigators record information on the number of hours in prone, and the number of days in prone position per patient. Additionally the following data is recorded: a) the predominant position adopted by the patient, defined as the position in which the patient spent most h/day, i.e., prone, lateral or supine position; b) the average number of h/day in that position; and c) the number of days of exposure to said position for a period of ≥ 6 h/day (AW-PP).

The primary outcome is defined as the receipt of endotracheal intubation. The decision to intubate was based on the criteria of the attending health-care team. However, intubation is recommended for anyone meeting the following criteria: deterioration of neurologic status, hemodynamic instability, or if two or more of the following criteria were met: decline in oxygen saturation with SpO2 < 90% for more than 5 minutes (not explained by technical failures), lack of improvement in the signs of respiratory muscle fatigue, impossibility to control airway secretions and respiratory acidosis with log10 hydrogen ion concentration (pH) < 7.30 [9]. Secondary outcome: hospital mortality. Secondary clinical outcomes: ICU and hospital length of stay, time to endotracheal intubation, and severe complications related to AW-PP.

Statistical analysis. The dynamics of the pandemic and the number of patients admitted to ICUs cannot be predicted. As many patients as possible were consecutively recruited without a predefined sample size (estimated 600).

Descriptive statistics will be used to describe the baseline characteristics of the patients. Categorical data will be presented as absolute frequency (n) and percentage (%) and continuous data as mean ± standard deviation (SD) or median and interquartile range (IR), respectively, as appropriate. Categorical variables will be compared by chi-square test (with Yates correction) or Fisher's exact tests, as appropriate. Continuous quantitative variables will be compared using the unpaired t-test or the Mann-Whitney test for normally and non-normally distributed variables, respectively. Each test will be two-tailed and a value of p<0.05 will be considered statistically significant. All analyses will be performed with STATA version 15.1.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years, admitted to the ICU
* Confirmed diagnosis of COVID-19 (real-time PCR)
* Receiving HFNO for at least 4 hours. Patients received HFNO when any of the following criteria were present: peripheral oxygen saturation (SpO2) < 92% with oxygen > 4 liters/minute; increased work of breathing with use of accessory respiratory muscles, and a respiratory rate > 30/min; PaO2/FiO2ratio < 200 mmHg.

Exclusion Criteria:

* Patients with respiratory failure secondary to a different etiology,
* Decreased level of consciousness,
* Presence of shock requiring vasopressors,
* Immediate need for intubation.
* Use of positive-pressure ventilation prior to HFNO, and f) with do-not intubate orders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included patients older than 17 years admitted to the ICU with a confirmed diagnosis of COVID-19 (real-time PCR) and receiving HFNO for at least 4 hours. Patients received HFNO when any of the following criteria were present: a) peripheral oxygen saturation (SpO2) < 92% with oxygen > 4 liters/minute; b) increased work of breathing with use of accessory respiratory muscles, and a respiratory rate > 30/min; c) PaO2/FiO2ratio < 200 mmHg. Patients with respiratory failure secondary to a different etiology, decreased level of consciousness, presence of shock requiring vasopressors, immediate need for intubation, use of positive-pressure ventilation prior to HFNO, and with do-not intubate orders were excluded.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Endotracheal Intubation | Up to 4 weeks
  Requirement of endotracheal intubation according to the criteria of previous studies (9,10).

SECONDARY OUTCOMES:
In-hospital mortality. | Up to 24 weeks
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Mariano Esperatti, Mar del Plata, Buenos Aires, Argentina

REFERENCES:
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Karagiannidis C, Mostert C, Hentschker C, Voshaar T, Malzahn J, Schillinger G, Klauber J, Janssens U, Marx G, Weber-Carstens S, Kluge S, Pfeifer M, Grabenhenrich L, Welte T, Busse R. Case characteristics, resource use, and outcomes of 10 021 patients with COVID-19 admitted to 920 German hospitals: an observational study. Lancet Respir Med. 2020 Sep;8(9):853-862. doi: 10.1016/S2213-2600(20)30316-7. Epub 2020 Jul 28. PMID 32735842
- [Result] Ranzani OT, Bastos LSL, Gelli JGM, Marchesi JF, Baiao F, Hamacher S, Bozza FA. Characterisation of the first 250,000 hospital admissions for COVID-19 in Brazil: a retrospective analysis of nationwide data. Lancet Respir Med. 2021 Apr;9(4):407-418. doi: 10.1016/S2213-2600(20)30560-9. Epub 2021 Jan 15. PMID 33460571
- [Result] Tan W, Xu DY, Xu MJ, Wang ZF, Dai B, Li LL, Zhao HW, Wang W, Kang J. The efficacy and tolerance of prone positioning in non-intubation patients with acute hypoxemic respiratory failure and ARDS: a meta-analysis. Ther Adv Respir Dis. 2021 Jan-Dec;15:17534666211009407. doi: 10.1177/17534666211009407. PMID 33888007
- [Result] Ponnapa Reddy M, Subramaniam A, Afroz A, Billah B, Lim ZJ, Zubarev A, Blecher G, Tiruvoipati R, Ramanathan K, Wong SN, Brodie D, Fan E, Shekar K. Prone Positioning of Nonintubated Patients With Coronavirus Disease 2019-A Systematic Review and Meta-Analysis. Crit Care Med. 2021 Oct 1;49(10):e1001-e1014. doi: 10.1097/CCM.0000000000005086. PMID 33927120
- [Result] Cardona S, Downing J, Alfalasi R, Bzhilyanskaya V, Milzman D, Rehan M, Schwartz B, Yardi I, Yazdanpanah F, Tran QK. Intubation rate of patients with hypoxia due to COVID-19 treated with awake proning: A meta-analysis. Am J Emerg Med. 2021 May;43:88-96. doi: 10.1016/j.ajem.2021.01.058. Epub 2021 Jan 27. PMID 33550104
- [Result] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Result] Francone M, Iafrate F, Masci GM, Coco S, Cilia F, Manganaro L, Panebianco V, Andreoli C, Colaiacomo MC, Zingaropoli MA, Ciardi MR, Mastroianni CM, Pugliese F, Alessandri F, Turriziani O, Ricci P, Catalano C. Chest CT score in COVID-19 patients: correlation with disease severity and short-term prognosis. Eur Radiol. 2020 Dec;30(12):6808-6817. doi: 10.1007/s00330-020-07033-y. Epub 2020 Jul 4. PMID 32623505
- [Result] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Result] Grieco DL, Menga LS, Cesarano M, Rosa T, Spadaro S, Bitondo MM, Montomoli J, Falo G, Tonetti T, Cutuli SL, Pintaudi G, Tanzarella ES, Piervincenzi E, Bongiovanni F, Dell'Anna AM, Delle Cese L, Berardi C, Carelli S, Bocci MG, Montini L, Bello G, Natalini D, De Pascale G, Velardo M, Volta CA, Ranieri VM, Conti G, Maggiore SM, Antonelli M; COVID-ICU Gemelli Study Group. Effect of Helmet Noninvasive Ventilation vs High-Flow Nasal Oxygen on Days Free of Respiratory Support in Patients With COVID-19 and Moderate to Severe Hypoxemic Respiratory Failure: The HENIVOT Randomized Clinical Trial. JAMA. 2021 May 4;325(17):1731-1743. doi: 10.1001/jama.2021.4682. PMID 33764378
- [Derived] Olmos M, Fuentes N, Busico M, Gallardo A, Vitali A, Costa ELV, Amato MBP, Bruhn A, Esperatti M; Argentine Collaborative Group on High Flow, Prone Positioning. Effectiveness of bundle of care on tolerance of awake-prone positioning in patients with acute respiratory failure. A multicenter observational study. Intensive Care Med. 2025 Feb;51(2):332-341. doi: 10.1007/s00134-025-07804-5. Epub 2025 Feb 17. PMID 39961842
- [Derived] Busico M, Fuentes NA, Gallardo A, Vitali A, Quintana J, Olmos M, Burns KEA, Esperatti M; Argentine Collaborative Group on High Flow and Prone Positioning. The Predictive Validity of the Berlin Definition of Acute Respiratory Distress Syndrome for Patients With COVID-19-Related Respiratory Failure Treated With High-Flow Nasal Oxygen: A Multicenter, Prospective Cohort Study. Crit Care Med. 2024 Jan 1;52(1):92-101. doi: 10.1097/CCM.0000000000006056. Epub 2023 Oct 16. PMID 37846935